CLINICAL TRIAL: NCT04031105
Title: Probing Homeostatic Plasticity With Priming Theta-burst Stimulation of the Dorsolateral Prefrontal Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Georg Kranz (Other)
Responsible Party: Sponsor-Investigator, Dr Georg Kranz, Principal Investigator, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PolyU 251002/19M
Record Dates: First submitted 2019-07-17; First posted 2019-07-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression Minor
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, single blind, parallel group experiment
Who Masked: Participant
Masking Description: Participants will not be told which arm they belong to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Condition 1 (Experimental): Priming sham TBS, followed by iTBS after an inter-stimulation-interval (ISI) of 0 minutes
  Interventions: Device: Theta-burst stimulation (TBS)
- Condition 2 (Experimental): Priming cTBS, followed by iTBS after an ISI of 0 minutes
  Interventions: Device: Theta-burst stimulation (TBS)
- Condition 3 (Experimental): Priming cTBS, followed by iTBS after an ISI of 10 minutes
  Interventions: Device: Theta-burst stimulation (TBS)
- Condition 4 (Experimental): Priming cTBS, followed by iTBS after an ISI of 20 minutes
  Interventions: Device: Theta-burst stimulation (TBS)

INTERVENTIONS:
Device: Theta-burst stimulation (TBS) — intermittent (iTBS) and continuous (cTBS) will be applied at an intensity of 70% or 100%* resting motor threshold (RMT) on the dorsolateral prefrontal cortex, position F3 (EEG 10-20 international system)
  *The optimal %RMT will be evaluated in a pilot study before commencement of the main study
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
Priming stimulation is a highly promising tool to boost the beneficial effects of therapeutic repetitive transcranial magnetic stimulation (rTMS) in psychiatry. The potentiating effects of priming stimulation, however, depend on the time interval between the priming and the test stimulation. Although it is known that too short and too long intervals have no effects, systematic studies that identify the time needed to maximize efficacy have not yet been done. Thus, there is a need for studies to investigate the effects of priming stimulation in order to fully utilize the potential benefits and advantages of this promising new rTMS protocol. This study will systematically investigate the neuromodulatory process underlying priming stimulation to enhance metaplasticity in the left dorsolateral prefrontal cortex (DLPFC) - one of the main targets for therapeutic rTMS - in individuals with subclinical depression.

The brain is a highly plastic organ and its activity can be influenced using rTMS. At the same time, the brain also has a mechanism - called homeostatic metaplasticity - which counteracts extreme plastic changes. Homeostatic metaplasticity therefore can limit the beneficial effects of brain stimulation interventions. However, priming stimulation protocols that include both a priming and a test stimulation session may utilize homeostatic metaplasticity to increase the beneficial effects of brain stimulation, although the optimal treatment parameters for priming are not known. Moreover, little is known about homeostatic metaplasticity in the DLPFC, an area that is particularly relevant for psychiatric conditions given its role in the top-down control of emotions. Here, the investigators will systematically study metaplasticity using priming theta-burst stimulation (TBS), a potent form of rTMS in the left DLPFC. Changes in blood oxygenation that signal brain activity changes will be assessed using functional near-infrared spectroscopy (fNIRS) at rest and during engagement in several cognitive tasks. The findings from this study will (1) elucidate the optimal time interval between priming and test stimulation; (2) elucidate the influence of priming TBS on emotion discrimination as well as executive function and its underlying brain activity in subclinical depression; and (3) validate homeostatic metaplasticity in the left DLPFC.

DETAILED DESCRIPTION:
No detailed description

ELIGIBILITY:
Inclusion Criteria:

1. age 18-35
2. education level of primary six or above
3. right-handedness
4. normal or corrected-to-normal vision
5. being able to understand the verbal instructions
6. willingness to sign the informed consent form

Exclusion Criteria:

1. a history of seizures
2. current or past psychiatric disorders
3. current or past severe internal or neurological illness
4. ferromagnetic implants <20cm from the head, cardiac pacemaker, deep brain stimulation and other common TMS exclusion criteria
5. history of substance dependence or abuse within the last 3 months
6. intake of any medication known to affect the excitation threshold (i.e., benzodiazepines, anticonvulsants).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin concentrations (Hb) during rest | Change from baseline Hb at 15 minutes post-stimulation
  Oxy- and deoxy-hemoglobin (HbO, HHb) and total Hb will be acquired using functional near-infrared spectroscopy (fNIRS)
Change in hemoglobin concentrations (Hb) while participants perform an emotion stroop task and verbal fluency task | Change from baseline Hb at 15 minutes after stimulation
  Oxy- and deoxy-hemoglobin (HbO, HHb) and total Hb will be acquired using functional near-infrared spectroscopy (fNIRS)

SECONDARY OUTCOMES:
Change in reaction time during emotion stroop task | Change from baseline reaction times at 15 minutes after stimulation
  Before and after stimulation, participants will perform a emotion stroop task. Participants are asked to indicate by button press in which color (red, yellow, blue, green) the word is presented on a computer screen,("c" for red, "v" for yellow, "n" for blue, "m" for green) . The total number and the reaction time of correct response will be recorded.
Change in the number of correctly responded colored words in the emotional Stroop task and correctly generated words in the verbal fluency task. | Change from baseline score at 15 minutes after stimulation
  Before and after stimulation, participants will perform an emotional Stroop task as described in Outcome 3. In addition, participants will also perform a verbal fluency task, In this task, participants are required to speak out as many unique words as possible during the word generation blocks, according to a given category (for example, name animals). The category will be presented at the center of the screen. The total number of correct answers will be recorded
Change in the number of correctly recognized emotion | Change from baseline score at 15 minutes after stimulation
  In addition, participants will perform an emotion-recognition accuracy task. They will be presented with 64 facial stimuli, consisting of sets of 16 sad, happy, fearful and neutral faces, in a randomized order. Faces will be presented for a maximum of 6s. Participants have to indicate the depicted emotion by button press (choice between 4 answers) within the presentation period.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Sharing upon request

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT04031105/Prot_SAP_002.pdf
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT04031105/ICF_003.pdf